CLINICAL TRIAL: NCT03590288
Title: Dynamic Monitor of Portacaval Pressure Gradient and Its Prognostic Value in Predicting Outcomes in Patients Undergoing TIPS
Brief Title: Dynamic Monitor of Portacaval Pressure Gradient
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Head of Department of Digestive Interventional Radiology, Air Force Military Medical University, China
Other Study IDs: PRESSURE GRADIENT MONITOR
Record Dates: First submitted 2018-06-28; First posted 2018-07-18 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2022-07

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis; Transjugular intrahepatic portosystemic shunt; Pressure gradient; Outcome prediction
MeSH Terms: conditions — Liver Cirrhosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TIPS group: Pressure gradient were measured in consecutive cirrhotic patients undergoing TIPS.
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt — Covered stents will be used, that will be dilated to 8 mm. The aim will be to reduce the portacaval pressure gradient (PPG) below to 25-75% of baseline. Not paralleled TIPS or over-dilatation are allowed.
  Embolisation, either with coils or bucrylate, can be performed, if it is felt necessary, especially in patients where portography shows the filling of big portosystemic collaterals feeding the varices.
  After TIPS, anticoagulation will not be used as a rule, but is allowed if the attending physician thinks that it is warranted.
  Measurement of portacaval pressure gradient will be done immediate after TIPS, then repeated 1-3 days and at 1 month after the procedure.
  A TIPS revision will be performed once shunt dysfunction is suspected.

SUMMARY:
Portacaval pressure gradient (PPG) plays an important role in prediction the outcomes of cirrhotic patients undergoing TIPS. An PPG over 20 mmHg indicates a high risk of failure to control bleeding or preventing rebleeding, while patients with PPG <12 mmHg are free from the risk of variceal bleeding. Transjugular intrahepatic portosystemic shunt (TIPS) markedly reduces PPG and is a very effective treatment for portal hypertension. A recent study showed that timing affects measurement of portacaval pressure gradient (PPG) after TIPS placement in patients with portal hypertension. The immediate PPG after TIPS placement cannot predict the long-term prognosis, while PPG measured with the patient on stable clinical conditions correlates with long term PPG and clinical outcomes. However, this finding remain to be validated. Previous studies have demonstrated that the achievement of a hepatic vein pressure gradient <12 mmHg eliminated the risk of recurrent variceal hemorrhage. Therefore, a post- TIPS PPG <12 mmHg was initially proposed as a hemodynamic target of TIPS, independent of the indication. It is important to note that most studies on hemodynamic targets were done before the introduction of covered stents and have not been adequately updated since then.Therefore, whether a post-TIPS PPG target <12 mmHg is the best cutoff for patients receiving a covered stent for the treatment of portal hypertension complications needs confirmation in well-designed studies.This study aims to dynamically monitor the change of PPG after TIPS procedure in patients with portal hypertension, and investigate its prognostic value in predicting patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with portal hypertensive complications
* Receiving TIPS due to variceal bleeding or refractory ascites
* Successful covered TIPS procedure
* Written informed consent

Exclusion Criteria:

* Lactating or pregnant
* Malignancies
* Uncontrolled infection (> grade 2)
* Severe cardiac, pulmonary or renal dysfunction
* Previously treated with TIPS
* Previous liver transplantation
* History of spontaneous overt HE or recurrent HE

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive cohort meeting the abovementioned criteria
Sampling Method: Non-Probability Sample
Enrollment: 567 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change of portacaval pressure gradient | The change of PPG from immediately to 1 month after the procedure
  The portacaval pressure gradient is the difference between the portal vein and the inferior vena cava pressures during portal angiography

SECONDARY OUTCOMES:
Portal hypertension related complications | 3 years
  The incidence of portal hypertensionrelated bleeding or ascites
Other portal hypertension complications | 3 years
  Spontaneous bacterial peritonitis, hepatorenal syndrome.
Hepatic encephalopathy | 3 years
  Hepatic encephalopathy
Survivial | 3 years
  Time from the procedure to the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lv Y, Wang Q, Luo B, Bai W, Li M, Li K, Wang Z, Xia D, Guo W, Li X, Yuan J, Zhang N, Wang X, Xie H, Pan Y, Nie Y, Yin Z, Fan D, Han G. Identifying the optimal measurement timing and hemodynamic targets of portal pressure gradient after TIPS in patients with cirrhosis and variceal bleeding. J Hepatol. 2025 Feb;82(2):245-257. doi: 10.1016/j.jhep.2024.08.007. Epub 2024 Aug 22. PMID 39181214